CLINICAL TRIAL: NCT05014880
Title: Impact of Time Restricted Eating on Exercise Capacity, Cardiometabolic Parameters, and Trimethylamine N-oxide (TMAO) Levels in Patients With Coronary Artery Disease (CAD) Undergoing Cardiac Rehabilitation
Brief Title: Impact of Time Restricted Eating on Patients With Coronary Artery Disease (CAD) Undergoing Cardiac Rehabilitation
Acronym: TRE x ICR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Salk Institute for Biological Studies (Other); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Pam Taub, MD, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200530
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease
Keywords: Time Restricted Eating; Circadian Rhythm; Cardiac Rehabilitation
MeSH Terms: conditions — Coronary Artery Disease; Intermittent Fasting

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICR (Intensive Cardiac Rehabilitation) (Placebo Comparator): 20 patients will be randomly assigned to the standard of care group, which will receive the standard health and nutritional wellness guidelines that are required of UCSD's 9-week ICR program, referred to as the "ICR" group.
  Interventions: Behavioral: ICR (Intensive Cardiac Rehabilitation)
- ICR x TRE (Intensive Cardiac Rehabilitation x Time-Restricted Eating) (Experimental): 20 patients will be randomly assigned to the Time-Restricted Eating (TRE) group which will be asked to limit the number of hours they eat in a day to 10 hours in addition to receiving the standard of care health and nutritional wellness guidelines that are required of UCSD's 9-week ICR program, referred to as the "ICR x TRE" group.
  Interventions: Behavioral: ICR x TRE (Intensive Cardiac Rehabilitation x Time-Restricted Eating)

INTERVENTIONS:
Behavioral: ICR (Intensive Cardiac Rehabilitation) — Participants in this arm will not have to adopt a 10-hour eating window while taking part in UCSD's 9-week ICR program.
  Arms: ICR (Intensive Cardiac Rehabilitation)
Behavioral: ICR x TRE (Intensive Cardiac Rehabilitation x Time-Restricted Eating) — Participants in this arm will adhere to a daily, consistent 10-hour eating window while undergoing UCSD's 9-week ICR program to see if there is an improvement on cardiometabolic parameters.
  Arms: ICR x TRE (Intensive Cardiac Rehabilitation x Time-Restricted Eating)

SUMMARY:
The purpose of this study is to see if reducing the number of hours during which one eats each day will help reduce levels of LDL cholesterol and improve other markers of metabolic and cardiovascular health (i.e. blood sugar levels and blood pressure). The study also aims to assess changes in exercise capacity and trimethylamine N-oxide (TMAO) levels in response to Time Restricted Eating (TRE) and Intensive Cardiac Rehabilitation (ICR) versus ICR alone. TMAO is a metabolite, or a substance, produced during digestion and metabolism. Preliminary data illustrates a correlation between high levels of TMAO and higher risk of cardiovascular disease and mortality. We will also be looking at participants' long-term cardiovascular health status after they complete the ICR program.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years
2. Enrollment and planned participation in UC San Diego's 9-week Intensive Cardiac Rehabilitation Program
3. Established diagnosis of coronary artery disease (concomitant systolic or diastolic HF is allowable)
4. Own a smartphone (Apple iOS or Android OS)
5. If patients are on cardiovascular medications (HMG CoA reductase inhibitors (statins), other lipid modifying drugs (including over the counter drugs such as red yeast rice and fish oil), anti-hypertensive, anti-diabetes drugs, no dose adjustments will be allowed during the study period.

Exclusion Criteria:

1. Taking insulin within the last 6 months.
2. Known inflammatory and/or rheumatologic disease.
3. Active tobacco abuse or illicit drug use or history of treatment for alcohol abuse.
4. Pregnant or breast-feeding women.
5. Shift workers with variable (e.g. nocturnal) hours.
6. Caregivers for dependents requiring frequent nocturnal care/sleep interruptions.
7. Planned international travel during study period.
8. Systolic HF alone.
9. Heart transplant within the past 1 year.
10. Presence of left ventricular assist device.
11. Uncontrolled arrhythmia (i.e. rate-controlled atrial fibrillation/atrial flutter are not exclusion criteria).
12. History of thyroid disease requiring dose titration of thyroid replacement medication(s) within the past 3 months (i.e. hypothyroidism on a stable dose of thyroid replacement therapy is not an exclusion).
13. History of adrenal disease.
14. History of malignancy undergoing active treatment, except non-melanoma skin cancer.
15. History of type I diabetes with ongoing insulin dependence.
16. History of eating disorders.
17. History of cirrhosis.
18. History of stage 4 or 5 chronic kidney disease or requiring dialysis.
19. History of HIV/AIDS.
20. Currently enrolled in a weight-loss or weight-management program. This does not include UC San Diego's Cardiac Rehabilitation Programs.
21. On a special or prescribed diet for other reasons (e.g. Celiac disease).
22. Currently taking any medication that is meant for, or has a known effect on, appetite.
23. Any history of surgical intervention for weight management.
24. Uncontrolled psychiatric disorder (including history of hospitalization for psychiatric illness).
25. Baseline eating window <14 hours per day as documented on mCC app.
26. Failure to use the smartphone app for documentation (defined as <2 meals/day for ≥3 days during baseline).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Exercise Capacity (MetS) | Baseline and Week 1-9
  Exercise Capacity

SECONDARY OUTCOMES:
Change in LDL cholesterol | Baseline and Week 9
  LDL cholesterol (mg/dL)
Change in non-HDL cholesterol | Baseline and Week 9
  non-HDL cholesterol (mg/dL)
Change in Triglycerides | Baseline and Week 9
  Triglycerides (mg/dL)

OTHER OUTCOMES:
Change in TMAO levels | Baseline and Week 9
  TMAO levels (uM)

CONTACTS AND LOCATIONS:
Overall Officials: Pam R Taub, MD, Principal Investigator — UC San Diego Health
Locations (1):
- Altman Clinical and Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided